CLINICAL TRIAL: NCT05483244
Title: Weaning Success in Different Weaning Strategies in Early Neurological Rehabilitation Patients - a Matched-pair Analysis
Status: Completed | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: Weaning Strategy
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Disorder; Respiratory Insufficiency
Keywords: early neurological rehabilitation; weaning strategy; weaning success
MeSH Terms: conditions — Nervous System Diseases; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- discontinuous weaning group: Patients of the discontinuous weaning group were disconnected from the respirator during the spontaneous breathing phases which could then take place via taken directly to the heat moist exchanger, high-flow therapy and/or speaking valve without pressure support by the respirator.
  Interventions: Other: discontinuous weaning
- continuous weaning group: In the case of continuous weaning, spontaneous breathing trial was supported by the respirator, but the positive endexpiratory pressure was lowered to an individual level (between 5 and 10 mbar) resulting in very little pressure support.
  Interventions: Other: continuous weaning

INTERVENTIONS:
Other: discontinuous weaning — Each day, a respiratory therapist evaluated whether a spontaneous breathing trial could be performed. Patients of the discontinuous weaning group were disconnected from the respirator during the spontaneous breathing phases which could then take place via heat moist exchanger, high-flow therapy and/or speaking valve without pressure support by the respirator (spontaneous breathing trial with heat moist exchanger).
  Heart rate, respiratory rate, blood pressure and mental condition of the patient (i. e. stress, fear) were monitored carefully for five to ten minutes and the Rapid Shallow Breathing Index was calculated. If the patient could keep the Rapid Shallow Breathing Index stable under 105/min/l (without a significant increase) over five minutes, the spontaneous breathing trial was regarded as successful and the weaning could be started. The duration of spontaneous breathing trial was extended according to the individual situation of the patient.
  Groups: discontinuous weaning group
Other: continuous weaning — Each day, a respiratory therapist evaluated whether a spontaneous breathing trial could be performed. In the case of continuous weaning, spontaneous breathing trial was supported by the respirator, but the positive endexpiratory pressure was lowered to an individual level (between 5 and 10 mbar) resulting in very little pressure support (spontaneous breathing trial trial under continuous positive airway pressure condition).
  Heart rate, respiratory rate, blood pressure and mental condition of the patient (i. e. stress, fear) were monitored carefully for five to ten minutes and the Rapid Shallow Breathing Index was calculated. If the patient could keep the Rapid Shallow Breathing Index stable under 105/min/l (without a significant increase) over five minutes, the spontaneous breathing trial was regarded as successful and the weaning could be started. The duration of spontaneous breathing trial was extended according to the individual situation of the patient.
  Groups: continuous weaning group

SUMMARY:
To enable weaning from mechanical ventilation, two different strategies may be distinguished: continuous weaning and discontinuous weaning. There is a lack of evidence of the superiority of one of both strategies is currently weak among early neurological rehabilitation patients. To the best of our knowledge, only one study including stroke patients compared different weaning strategies and showed a significantly shorter duration of mechanical ventilation during continuous than during discontinuous weaning, which is in contrast to the results of the largest weaning study with patients on medical-surgical intensive care units. In addition, further inconsistent results were reported from studies with chronic obstructive pulmonary disease patients, which might be due to disease duration and/or duration of prior mechanical ventilation in the acute care hospital.

This small number of studies with controversial results indicates that there is a considerable need for further research. The current study intended to compare the rehabilitation outcome of early neurological rehabilitation patients, weaned by different strategies (continuous vs. discontinuous) through a matched-pair analysis.

DETAILED DESCRIPTION:
Early rehabilitation patients admitted in the year 2020 to the intensive care unit of the BDH-Clinic Hessisch Oldendorf were screened for continuous weaning strategy by a respiratory therapist, retrospectively. Selected patients and a matching patient with a continuous weaning strategy was then identified in the clinical database (years 2017 to 2020) to generate a matched-pair according to the following characteristics: age, gender, diagnosis and severity of disease (early rehabilitation barthel index upon admission).

All data was collected retrospectively. Pre-existing diseases, disease duration (days between onset of neurological disease and admission to early neurological rehabilitation facility) and duration of mechanical ventilation before admission to early neurological rehabilitation facility were collected from medical records of the referring hospital. The course of weaning was described by the duration of mechanical ventilation (total hours and number of days), the weaning success and the removal of tracheal cannula. In addition, further information ( length of stay, the duration and time point of the first spontanous breathing trial as well as the occurrence of adverse events during rehabilitation) was documented for every patient.

Data was analyzed by the Statistical Package for Social Sciences (SPSS; version 26). Descriptive statistics were done and presented as median and interquartile range (IQR, 25th and 75th percentiles). For categorical data, descriptive statistics were calculated as frequencies. Differences between groups (continuous vs. discontinuous weaning) were analyzed by Mann-Whitney U test or Chi²-Test. Correlation analyses were performed by Spearman. A p-value <0.05 was considered as stastical significant.

ELIGIBILITY:
Inclusion Criteria (continuous weaning group):

* mechanical ventilation at admission to neurological rehabilitation
* weaned by a continuous or discontinuous weaning strategy

Exclusion Criteria:

* pre-existing mechanical ventilation before disease onset
* mixed weaning strategies (continuous and discontinuous) during weaning process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neurological main diagnoses, who admitted to early neurological rehabilitation and are under mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
weaning success | through study completion, an average of 70 days
  number of patients who could weaned sucessfully from mechanical ventilation

SECONDARY OUTCOMES:
weaning duration | through study completion, an average of 70 days
  duration of mechnaical ventilation (in hours)

CONTACTS AND LOCATIONS:
Overall Officials: Simone B Schmidt, Dr., Principal Investigator — BDH-Klinik Hessisch Oldendorf
Locations (1):
- Institute for Neurorehabilitation Research, BDH-Clinic Hessich Oldendorf, Hessisch Oldendorf, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Background] Teismann IK, Oelschlager C, Werstler N, Korsukewitz C, Minnerup J, Ringelstein EB, Dziewas R. Discontinuous versus Continuous Weaning in Stroke Patients. Cerebrovasc Dis. 2015;39(5-6):269-77. doi: 10.1159/000381222. Epub 2015 Apr 8. PMID 25871403
- [Background] Vitacca M, Vianello A, Colombo D, Clini E, Porta R, Bianchi L, Arcaro G, Vitale G, Guffanti E, Lo Coco A, Ambrosino N. Comparison of two methods for weaning patients with chronic obstructive pulmonary disease requiring mechanical ventilation for more than 15 days. Am J Respir Crit Care Med. 2001 Jul 15;164(2):225-30. doi: 10.1164/ajrccm.164.2.2008160. PMID 11463592
- [Background] Matic I, Danic D, Majeric-Kogler V, Jurjevic M, Mirkovic I, Mrzljak Vucinic N. Chronic obstructive pulmonary disease and weaning of difficult-to-wean patients from mechanical ventilation: randomized prospective study. Croat Med J. 2007 Feb;48(1):51-8. PMID 17309139